CLINICAL TRIAL: NCT00294216
Title: A Double Blind Comparison of Omacor and Placebo in Patients Awaiting Endarterectomy to Investigate the Effect on Carotid Plaque Stability
Brief Title: Omacor and Placebo in Carotid Plaque Stability
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pronova BioPharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CTN K85 02025
Record Dates: First submitted 2006-02-17; First posted 2006-02-20 (Estimated); Last update posted 2006-02-20 (Estimated); Status verified 2006-02

CONDITIONS: Cardiovascular Disease
Keywords: Omacor; Omega-3 PUFA; Endarterectomy; Carotid Plaque stability; Structural changes; inflammation
MeSH Terms: conditions — Cardiovascular Diseases; Inflammation | interventions — Fatty Acids, Omega-3

INTERVENTIONS:
Drug: Omega-3-acid ethyl ester 90 (n-3 PUFA)

SUMMARY:
The purpose of this study is to investigate the effect of intake of Omacor (Omega-3-acid ethyl ester 90) 2g/day on specified parameters related to the stability of carotid plaque in patients awaiting endarterectomy.

DETAILED DESCRIPTION:
There is evidence both from epidemiological studies and large clinical trials that consumption of long-chain Omega-3 polyunsaturated fatty acids (PUFA) found in oily fish and fish oils, protects against cardiovascular disease in Western Populations. The large clinical trial GISSI-Prevention showed radical reductions in Cardiovascular Disease and Sudden Cardiac Death after the intake of Omega-3 PUFA, and statistically significant effects were seen after only a few months of use.

One of the models for explaining this markedly effect hypothesizes that Omega-3 PUFA, with its anti inflammatory effects, might act to stabilize atherosclerotic plaques by decreasing infiltration of inflammatory cells into the plaques and/or by decreasing the activity of these cells once resident in the plaque. A previous clinical study has showed increased incorporation of the Omega-3 fatty acids EPA and DHA in carotid plaque after intake of Omega-3 PUFA. The morphological properties of the plaque was also altered, showing thicker fibrous caps and less inflammation determined by the AHA and modified AHA classification.

These findings are important to confirm. Secondly additional indicators of plaque stability are required to strengthen the hypothesis. Also the mechanisms by which the morphological changes come about need to be identified. The model that is being used assesses structural changes associated with plaque rupture and instability through different important variables.

Comparisons: Double blind comparison of Omacor 2g/day and placebo in patients awaiting endarterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Males of females above 18 years of age
* Patients awaiting carotid endarterectomy
* Written Informed Consent

Exclusion Criteria:

* Patients consuming fish oil or evening primrose oil preparations
* Patients eating > 2 oily fish meals per week
* Patients requiring operation within 7 days
* Pregnant or breastfeeding
* Patients participating in other clinical studies involving treatment with drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121
Dates: Start 2003-08; Study Completion 2005-07

PRIMARY OUTCOMES:
The primary objective is to compare the carotid plaque stability after placebo versus Omega-3 fatty acid treatment by assessing structural changes associated with plaque rupture and instability. The composite endpoint includes changes in
(1) the size of the lipid pool,
(2) the number of foam cells,
(3) the presence of haemorrhage,
(4) the number of macrophages in lesions and
(5) the overall density of inflammation in the plaque as a whole and
(6) in fibrous caps of lesions.

SECONDARY OUTCOMES:
(1) the size of the lipid pool,
(2) the number of foam cells,
(3) the presence of haemorrhage,
(4) the number of macrophages in lesions and
(5) the overall density of inflammation in the plaque as a whole and
(6) in fibrous caps of lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Philip C. Calder, PhD, Principal Investigator — University of Southampton, School of Medicine, Institute of Human Nutrition
Locations (1):
- University of Southampton, School of medicine, Southampton, United Kingdom

REFERENCES:
- [Background] Thies F, Garry JM, Yaqoob P, Rerkasem K, Williams J, Shearman CP, Gallagher PJ, Calder PC, Grimble RF. Association of n-3 polyunsaturated fatty acids with stability of atherosclerotic plaques: a randomised controlled trial. Lancet. 2003 Feb 8;361(9356):477-85. doi: 10.1016/S0140-6736(03)12468-3. PMID 12583947
- [Derived] Cawood AL, Ding R, Napper FL, Young RH, Williams JA, Ward MJ, Gudmundsen O, Vige R, Payne SP, Ye S, Shearman CP, Gallagher PJ, Grimble RF, Calder PC. Eicosapentaenoic acid (EPA) from highly concentrated n-3 fatty acid ethyl esters is incorporated into advanced atherosclerotic plaques and higher plaque EPA is associated with decreased plaque inflammation and increased stability. Atherosclerosis. 2010 Sep;212(1):252-9. doi: 10.1016/j.atherosclerosis.2010.05.022. Epub 2010 May 20. PMID 20542512